CLINICAL TRIAL: NCT05915793
Title: Combined Effects of Diaphragm Strengthening and Accessory Muscles Stretchings in Asthma Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: REC/RCR&AHS/23/0315
Record Dates: First submitted 2023-06-14; First posted 2023-06-23 (Actual); Last update posted 2023-06-23 (Actual); Status verified 2023-06

CONDITIONS: Asthma
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Diaphragm strengthening and accessory muscles stretchings (Experimental)
  Interventions: Other: Diaphragm strengthening and accessory muscles stretchings
- Diaphragm strengthening (Active Comparator)
  Interventions: Other: Diaphragm strengthening

INTERVENTIONS:
Other: Diaphragm strengthening and accessory muscles stretchings — Diaphragm strengthening and accessory muscles stretchings
  Arms: Diaphragm strengthening and accessory muscles stretchings
Other: Diaphragm strengthening — Diaphragm strengthening
  Arms: Diaphragm strengthening

SUMMARY:
Asthma is a multifactorial and chronic inflammatory disease in older patients affecting many people worldwide with high cost of pharmacological treatment and physiotherapy interventions. It is characterized by a variety of symptoms including airway inflammation, bronchial hyper-responsiveness, and transient and reversible airway obstruction. Typical clinical features include wheezing, coughing, resting and/or exertional dyspnea, and chest tightness. Lung hyperinflation affects ability to inspire and increases the work of breathing.

Long and short acting corticosteroids and leukotriene are considered effective pharmacological interventions while inspiratory muscle training, incentive spirometry, purse lip breathing, and diaphragm strengthening are considered effective physiotherapy interventions for asthma patients. To find the combined effects of diaphragm strengthening and accessory muscle stretching on chest expansion, pulmonary function, dyspnea and exercise capacity in asthmatic patients. A randomized controlled trial will be conducted at Gulab Davi teaching Hospital Lahore through convenient sampling technique on 40 patients which will be allocated through concealed opaque envelop into Group A and Group Pretreatment values of pulmonary function and chest expansion will be recorded. And patient's perception of exertion through Modified Borg's rating of perceived exertion (RPE) and HRQOL for quality of life will be assessed before and after treatment. Group A will be treated with diaphragm strengthening and Group B will be treated with diaphragm strengthening and accessory muscles stretching. Treatment evaluation will be done after 4 weeks. Data will be analyzed using SPSS software version 25. After assessing normality of data by Shapiro-Wilk test, it will be decided either parametric or non-parametric test will be use within a group or between two groups.

ELIGIBILITY:
Inclusion Criteria:

* Age group of 40-65 years
* Both male and females
* Phase-2 asthma patients
* Patients hemodynamically stable

Exclusion Criteria:

* Patients having pulmonary tumors
* Patients of Having cough and sputum
* Patients having TB and emphysema
* Patients with pneumonia, pneumonectomy or other lungs surgical procedures

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Estimated)
Dates: Start 2023-02-01 (Actual); Primary Completion 2023-08-29 (Estimated); Study Completion 2023-08-29 (Estimated)

PRIMARY OUTCOMES:
Modified Borg scale of exertion | 6 weeks
  The Modified Borg Dyspnea Scale (MBS) is a 0 to 10 rated numerical score used to measure dyspnea as reported by the patient during submaximal exercise and is routinely administered during six-minute walk testing (6MWT)
6 MWT | 6 weeks
  The 6MWT was used to detect participants' functional capacity by measuring the distance they traveled during the walk test. For the 6MWT assessment, the participants were encouraged to walk as far as they could during 6 min over a flat 100-feet surface, and for consistency, the researchers used constant verbal cues and positive feedback to encourage the participants to complete the task

SECONDARY OUTCOMES:
Quality of life questionnaire | 6 weeks
  HRQOL is one of several variables commonly studied in the field of medical outcomes research. It encompasses a wide range of human experience, including functioning and subjective responses to illness. Contemporary interpretations of HRQOL are based on the World Health Organization's definition of health as a state of complete physical, mental, and social well-being and not merely the absence of disease. contemporary HRQOL instrument domains are scored with a range of 0-100, with higher values representing better outcomes.
  To make useful inferences regarding absolute scores or change scores over time, it is important to determine what meaning different numerical values have. When no such thresholds have been established, one can roughly approximate the smallest difference that is important to the patient as one-third to one-half of a standard deviation

CONTACTS AND LOCATIONS:
Overall Officials: Ameena Amjad, tDPT, Principal Investigator — Riphah International University
Locations (1):
- Gulab Devi Hospital, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Gomieiro LT, Nascimento A, Tanno LK, Agondi R, Kalil J, Giavina-Bianchi P. Respiratory exercise program for elderly individuals with asthma. Clinics (Sao Paulo). 2011;66(7):1163-9. doi: 10.1590/s1807-59322011000700007. PMID 21876968
- [Background] Worldwide variation in prevalence of symptoms of asthma, allergic rhinoconjunctivitis, and atopic eczema: ISAAC. The International Study of Asthma and Allergies in Childhood (ISAAC) Steering Committee. Lancet. 1998 Apr 25;351(9111):1225-32. PMID 9643741
- [Background] Bradshaw D, Groenewald P, Laubscher R, Nannan N, Nojilana B, Norman R, Pieterse D, Schneider M, Bourne DE, Timaeus IM, Dorrington R, Johnson L. Initial burden of disease estimates for South Africa, 2000. S Afr Med J. 2003 Sep;93(9):682-8. PMID 14635557
- [Background] GBD 2015 Chronic Respiratory Disease Collaborators. Global, regional, and national deaths, prevalence, disability-adjusted life years, and years lived with disability for chronic obstructive pulmonary disease and asthma, 1990-2015: a systematic analysis for the Global Burden of Disease Study 2015. Lancet Respir Med. 2017 Sep;5(9):691-706. doi: 10.1016/S2213-2600(17)30293-X. Epub 2017 Aug 16. PMID 28822787
- [Background] Asher I, Pearce N. Global burden of asthma among children. Int J Tuberc Lung Dis. 2014 Nov;18(11):1269-78. doi: 10.5588/ijtld.14.0170. PMID 25299857
- [Background] Burney P, Jarvis D, Perez-Padilla R. The global burden of chronic respiratory disease in adults. Int J Tuberc Lung Dis. 2015 Jan;19(1):10-20. doi: 10.5588/ijtld.14.0446. PMID 25519785
- [Background] Hasnain SM, Khan M, Saleem A, Waqar MA. Prevalence of asthma and allergic rhinitis among school children of Karachi, Pakistan, 2007. J Asthma. 2009 Feb;46(1):86-90. doi: 10.1080/02770900802513023. PMID 19191144
- [Background] Arm JP, Horton CE, Mencia-Huerta JM, House F, Eiser NM, Clark TJ, Spur BW, Lee TH. Effect of dietary supplementation with fish oil lipids on mild asthma. Thorax. 1988 Feb;43(2):84-92. doi: 10.1136/thx.43.2.84. PMID 3353893
- [Background] Weiler JM. Exercise-induced asthma: a practical guide to definitions, diagnosis, prevalence, and treatment. Allergy Asthma Proc. 1996 Nov-Dec;17(6):315-25. doi: 10.2500/108854196778606437. PMID 8993724
- [Background] Boulet LP, Becker A, Berube D, Beveridge R, Ernst P. Canadian Asthma Consensus Report, 1999. Canadian Asthma Consensus Group. CMAJ. 1999 Nov 30;161(11 Suppl):S1-61. PMID 10906907
- [Background] Barnes PJ. The cytokine network in asthma and chronic obstructive pulmonary disease. J Clin Invest. 2008 Nov;118(11):3546-56. doi: 10.1172/JCI36130. PMID 18982161
- [Background] Barnes PJ. Immunology of asthma and chronic obstructive pulmonary disease. Nat Rev Immunol. 2008 Mar;8(3):183-92. doi: 10.1038/nri2254. Epub 2008 Feb 15. PMID 18274560
- [Background] Hallstrand TS, Debley JS, Farin FM, Henderson WR Jr. Role of MUC5AC in the pathogenesis of exercise-induced bronchoconstriction. J Allergy Clin Immunol. 2007 May;119(5):1092-8. doi: 10.1016/j.jaci.2007.01.005. Epub 2007 Feb 26. PMID 17321575
- [Background] Reid WD, Dechman G. Considerations when testing and training the respiratory muscles. Phys Ther. 1995 Nov;75(11):971-82. doi: 10.1093/ptj/75.11.971. PMID 7480127
- [Background] Deesomchok A, Fisher T, Webb KA, Ora J, Lam YM, Lougheed MD, O'Donnell DE. Effects of obesity on perceptual and mechanical responses to bronchoconstriction in asthma. Am J Respir Crit Care Med. 2010 Jan 15;181(2):125-33. doi: 10.1164/rccm.200906-0934OC. Epub 2009 Nov 12. PMID 19910609
- [Background] Illi SK, Held U, Frank I, Spengler CM. Effect of respiratory muscle training on exercise performance in healthy individuals: a systematic review and meta-analysis. Sports Med. 2012 Aug 1;42(8):707-24. doi: 10.1007/BF03262290. PMID 22765281
- [Background] Turner LA, Mickleborough TD, McConnell AK, Stager JM, Tecklenburg-Lund S, Lindley MR. Effect of inspiratory muscle training on exercise tolerance in asthmatic individuals. Med Sci Sports Exerc. 2011 Nov;43(11):2031-8. doi: 10.1249/MSS.0b013e31821f4090. PMID 21502887
- [Background] Hallstrand TS, Bates PW, Schoene RB. Aerobic conditioning in mild asthma decreases the hyperpnea of exercise and improves exercise and ventilatory capacity. Chest. 2000 Nov;118(5):1460-9. doi: 10.1378/chest.118.5.1460. PMID 11083702
- [Background] Lucas SR, Platts-Mills TA. Physical activity and exercise in asthma: relevance to etiology and treatment. J Allergy Clin Immunol. 2005 May;115(5):928-34. doi: 10.1016/j.jaci.2005.01.033. PMID 15867847
- [Background] Boyd A, Yang CT, Estell K, Ms CT, Gerald LB, Dransfield M, Bamman M, Bonner J, Atkinson TP, Schwiebert LM. Feasibility of exercising adults with asthma: a randomized pilot study. Allergy Asthma Clin Immunol. 2012 Aug 3;8(1):13. doi: 10.1186/1710-1492-8-13. PMID 22863207
- [Background] Westwood K, Griffin M, Roberts K, Williams M, Yoong K, Digger T. Incentive spirometry decreases respiratory complications following major abdominal surgery. Surgeon. 2007 Dec;5(6):339-42. doi: 10.1016/s1479-666x(07)80086-2. PMID 18080608
- [Background] Lotters F, van Tol B, Kwakkel G, Gosselink R. Effects of controlled inspiratory muscle training in patients with COPD: a meta-analysis. Eur Respir J. 2002 Sep;20(3):570-6. doi: 10.1183/09031936.02.00237402. PMID 12358330
- [Background] Chung Y, Huang TY, Liao YH, Kuo YC. 12-Week Inspiratory Muscle Training Improves Respiratory Muscle Strength in Adult Patients with Stable Asthma: A Randomized Controlled Trial. Int J Environ Res Public Health. 2021 Mar 22;18(6):3267. doi: 10.3390/ijerph18063267. PMID 33809922